CLINICAL TRIAL: NCT02474264
Title: The Link Between BRCA Mutation and Endothelial Function - A Pilot Study
Brief Title: The Link Between BRCA Mutation and Endothelial Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 0594-14-RMC
Record Dates: First submitted 2015-02-23; First posted 2015-06-17 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2016-10

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- male BRCA mutations carriers (Other): Endothelial function assessment and Cardiovascular biomarkers
  Interventions: Other: Endothelial function assessment; Other: Cardiovascular biomarkers; Other: Endothelial cells
- healthy males - control group (Other): Endothelial function assessment and Cardiovascular biomarkers
  Interventions: Other: Endothelial function assessment; Other: Cardiovascular biomarkers; Other: Endothelial cells

INTERVENTIONS:
Other: Endothelial function assessment — reactive hyperemia index
Other: Cardiovascular biomarkers — Cardiovascular biomarkers will be measure to test other aspects of endothelial and cardiac function: high-sensitivity troponin (hsTn) , C-reactive protein , D-dimer, N-terminal pro-brain natriuretic peptide (NT-proBNP)
Other: Endothelial cells — Endothelial Progenitor Cells and Circulating Endothelial Cells profiles- will be characterized to evaluate endothelial injury.

SUMMARY:
This study evaluates the effect of BRCA1&2 mutations on cardiovascular diseases by to comparing the endothelial function of male BRCA mutation carriers with that of age matched non-BRCA mutation carriers.

ELIGIBILITY:
Inclusion Criteria:

* Known carrier or non-carrier, confirmed by genetic testing of BRCA 1/2 mutation
* Able and willing to sign an informed consent

Exclusion Criteria:

* History of, or current, malignancy
* History of:

  * Myocardial infarction
  * Ischemic or Hemorrhagic cerebrovascular conditions
  * Arterial embolic and thrombotic events
  * Ischemic heart disease
  * Prior coronary artery or ilio-femoral artery revascularization (percutaneous or surgical procedures)
  * Peripheral vascular disease (e.g. claudication, prior vascular surgery/intervention)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
reactive hyperemia index will be assessed using the Endo-PAT2000 | at baseline
  will be assessed using the Endo-PAT2000

SECONDARY OUTCOMES:
The level of high sensitivity troponin (hsTn) - a cardiovascular risk biomarker will be measured | at baseline
  high sensitivity troponin (hsTn)
The level of C-reactive protein - a cardiovascular risk biomarker will be measured | at baseline
  C-reactive protein
The level of D-dimer - a cardiovascular risk biomarker will be measured | at baseline
  D-dimer
The level of N-terminal pro-brain natriuretic peptide (NT-proBNP) - a cardiovascular risk biomarker will be measured | at baseline
  N-terminal pro-brain natriuretic peptide (NT-proBNP)
Endothelial Progenitor Cells profile (EPC) - will be characterized to evaluate endothelial injury. | at baseline
  Endothelial Progenitor Cells (EPC)
Circulating Endothelial Cells profile (CEC) - will be characterized to evaluate endothelial injury. | at baseline
  Circulating Endothelial Cells (CEC)

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD, PhD, Principal Investigator — Rabn Medical Center, Beilinson Campus
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided